CLINICAL TRIAL: NCT06268444
Title: Infant Sleep and Exposure to Mixture of Environmental Pollutants
Brief Title: Infant Sleep and Exposure to Mixture of Chemical Environmental Pollutants
Acronym: SOLANGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PI2023_843_0077
Record Dates: First submitted 2024-02-13; First posted 2024-02-20 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Newborn; Chemical Pollutants Exposure; Sleep
Keywords: sleep; Newborn; chemical pollutants exposure
MeSH Terms: interventions — Milk, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- New born (Experimental)
  Interventions: Device: 7-day actimetry sleep recording; Other: Determination of environmental pollutants in breast milk; Other: Measurements of environmental pollutants in indoor air deposited on the bracelet worn by the child; Other: Continuous recording of the child's temperature for 7 days; Other: Use of a sleep diary for 7 days; Other: Parental questionnaire of environmental exposure

INTERVENTIONS:
Device: 7-day actimetry sleep recording — 7-day actimetry sleep recording
Other: Determination of environmental pollutants in breast milk — Determination of environmental pollutants in breast milk
Other: Measurements of environmental pollutants in indoor air deposited on the bracelet worn by the child — Measurements of environmental pollutants in indoor air deposited on the bracelet worn by the child
Other: Continuous recording of the child's temperature for 7 days — Continuous recording of the child's temperature for 7 days
Other: Use of a sleep diary for 7 days — Use of a sleep diary for 7 days
Other: Parental questionnaire of environmental exposure — Parental questionnaire of environmental exposure

SUMMARY:
During their first year of life, children spend more than half their time sleeping, a function essential to their neurodevelopment. This period of maturation and development of the future adult is considered extremely vulnerable to environmental exposure. During this period, the child's diet is mainly provided by breastfeeding, where persistent chemical substances have been found. A cocktail of 19 mostly persistent substances (POPs) present in breast milk has recently been identified as the main contributor to neurodevelopmental risk. However, the reality of their impact on neurophysiological development, in particular on infant sleep, has yet to be assessed.

In this project, the sleep of children under 6 months of age will be studied using an actimetry watch worn for 7 days by the child, accompanied by a sleep diary. Exposure to environmental pollutants will be assessed by measuring their presence in the infant's milk (breastfeeding) and wearing a silicone bracelet to collect air pollutants. A questionnaire on exposure will complement this evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Infant less than 6 months of age still on milk diet (total)

Exclusion Criteria:

* Infants with neurological or neurobehavioral disorders
* Families who wish to relocate within 7 days of inclusion
* Minor parents deprived of their parental rights, not understanding French, in a state of stress, overwhelmed or vulnerable.
* Non-affiliation to a social security system

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
total sleep time per day in infants using actimetry | 7 days
  total sleep time per day (min)) in infants using actimetry

SECONDARY OUTCOMES:
Concentration of various substances in breast milk | 1 day
concentration of chemical polluants on newborn bracelets | 1 day
Child Temperature level (°C) | 7 days

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France